CLINICAL TRIAL: NCT05346432
Title: Effects of Lactobacillus Paracasei PS23 on Anti-fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chi-Chang Huang (Other)
Collaborators: Bened Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Chi-Chang Huang, Principal Investigator, National Taiwan Sport University
Organization: National Taiwan Sport University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 22-003-A2
Record Dates: First submitted 2022-03-24; First posted 2022-04-26 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PS23 (Experimental): The PS23 belongs to Lactobacillus paracasei group, 2 caps daily use.
  Interventions: Dietary Supplement: PS23
- heat-treated PS23 (Experimental): PS23 heat-treated, 2 caps daily use.
  Interventions: Dietary Supplement: PS23
- placebo (Placebo Comparator): The placebo capsule contains microcrystalline cellulose, 2 caps daily use.
  Interventions: Dietary Supplement: PS23

INTERVENTIONS:
Dietary Supplement: PS23 — PS23 belongs to Lactobacillus paracasei group.Probiotic capsules contain 10 billion CFU (colony forming units) of PS23

SUMMARY:
This research is to explore the effects of supplementing Lactobacillus paracasei PS23 to reduce fatigue and improve physical fitness after exhaustive exercise.

DETAILED DESCRIPTION:
Studies have found that the intestinal flora of athletes is different from that of ordinary people, and short-chain fatty acids play a very important role. Previous animal experiments have found that supplementing with specific probiotics can slow down muscle loss in aging mice. In addition, clinical studies have found that supplementing with probiotics can improve sports performance by regulating the intestinal flora and related metabolites. Therefore, the purpose of this research is to explore the effects of supplementing Lactobacillus paracasei PS23 to reduce fatigue and improve physical fitness after exhaustive exercise. This study compares supplementary samples with placebo and adopts a double-blind study design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and women aged 20-40 who are generally non-athletic players

Exclusion Criteria:

* BMI≧27
* Known allergy to probiotics
* Have current or history of inflammatory bowel disease
* Patients using of other probiotic products (sachet, capsule or tablet) within the preceding two weeks
* Those who have taken medication such as anti-inflammatory pain killer or antibiotics in the past one month
* smoker and alcoholic
* Who have been injured within 6 months
* Who has been diagnosed and treated of cardiovascular disease, hypertension, metabolic disease, asthma, or cancer
* Have undergone surgery of liver, bladder, or gastrointestinal tract
* Who has conflict of interest with PI

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Stress assessment - difference of Testosterone level | From Baseline to 6 Weeks Assessed
  To assess inflammation indicators, volunteers fasted for at least 8 hours before performing muscle exhaustion exercises. At designated time points in the recovery period, including baseline (0) and 3h, 24h, and 48 after exercise, blood samples were collected with brachial venous catheters. Used commercial kit human Testosterone (Cayman, Mich, USA) and Elisa reader (PerkinElmer, Massachusetts, USA) for analysis Male 265-923 (in ng/dl) Female 15-70 (in ng/dl) for 19 years and older
Difference in Clinical Biochemistry of CK level | From Baseline to 6 Weeks Assessed, including baseline (0) and 3h, 24h, and 48 after exercise
  To assess inflammation indicators, volunteers fasted for at least 8 hours before performing muscle exhaustion exercises. At designated time points in the recovery period, blood samples were collected with brachial venous catheters. Assess serum CK(Creatine Kinase, U/L) to monitor physiological fitness. Serum CK (U/L), were assessed for monitoring physiological adaptation. All biochemical indices were assessed using an autoanalyzer (Hitachi 7060, Tokyo, Japan).
Difference of Muscle damage - blood level of myoglobin | From Baseline to 6 Weeks Assessed, including baseline (0) and 3h, 24h, and 48 after exercise
  To assess Muscle damage such as myoglobin (Female:14.3~65.8, Male:17.4~105.7) Volunteers fasted for at least 8 hours before performing muscle exhaustion exercises. At designated time points in the recovery period, blood samples were collected with brachial venous catheters. Used commercial kit human myoglobin (Cayman, Mich, USA) and Elisa reader (PerkinElmer, Massachusetts, USA) for analysis
Oxidative stress assessment - blood of MDA level | From Baseline to 6 Weeks Assessed
  comparing blood levels of oxidative markers such as Malondialdehyde (MDA)
Difference in Oxidative stress - blood level of CRP | From Baseline to 6 Weeks Assessed, including baseline (0) and 3h, 24h, and 48 after exercise
  To assess inflammation indicators, volunteers fasted for at least 8 hours before performing muscle exhaustion exercises. At designated time points in the recovery period, blood samples were collected with brachial venous catheters. Used commercial kit human CRP (Cayman, Mich, USA) and Elisa reader (PerkinElmer, Massachusetts, USA) for analysis
The Countermovement Jump (CMJ) Test | From Baseline to 6 Weeks Assessed, In this study, this assessment was performed before and 24 and 48h after the exhaustive exercise program.
  The CMJ test is a practical, effective, reliable, and simple method of measuring lower limb strength, which is related to the maximum speed, strength and explosive force of the lower limbs. For this test, participants stood on the Kistler force measurement platform (9260AA, Kistler Co., Ltd., Switzerland) on both feet and performed to inspection. During the test, they were asked to put their hands on their hips and remain on the platform. After that, they were asked to squat down until the knees bent 90 degrees and then to immediately jump as high as possible. The average power (MF), were recorded during the jump. Each participant repeated the test 3 times, and CMJ data were obtained at the designated points. The instrument was calibrated for each individual's weight.
The Countermovement Jump (CMJ) Test | From Baseline to 6 Weeks Assessed, In this study, this assessment was performed before and 24 and 48h after the exhaustive exercise program.
  The CMJ test is a practical, effective, reliable, and simple method of measuring lower limb strength, which is related to the maximum speed, strength and explosive force of the lower limbs. For this test, participants stood on the Kistler force measurement platform (9260AA, Kistler Co., Ltd., Switzerland) on both feet and performed to inspection. During the test, they were asked to put their hands on their hips and remain on the platform. After that, they were asked to squat down until the knees bent 90 degrees and then to immediately jump as high as possible. The peak power (Fpeak), were recorded during the jump. Each participant repeated the test 3 times, and CMJ data were obtained at the designated points. The instrument was calibrated for each individual's weight.
The Countermovement Jump (CMJ) Test | From Baseline to 6 Weeks Assessed, In this study, this assessment was performed before and 24 and 48h after the exhaustive exercise program.
  The CMJ test is a practical, effective, reliable, and simple method of measuring lower limb strength, which is related to the maximum speed, strength and explosive force of the lower limbs. For this test, participants stood on the Kistler force measurement platform (9260AA, Kistler Co., Ltd., Switzerland) on both feet and performed to inspection. During the test, they were asked to put their hands on their hips and remain on the platform. After that, they were asked to squat down until the knees bent 90 degrees and then to immediately jump as high as possible. flight time (FT) were recorded during the jump. Each participant repeated the test 3 times, and CMJ data were obtained at the designated points. The instrument was calibrated for each individual's weight.
The Countermovement Jump (CMJ) Test | From Baseline to 6 Weeks Assessed, In this study, this assessment was performed before and 24 and 48h after the exhaustive exercise program.
  The CMJ test is a practical, effective, reliable, and simple method of measuring lower limb strength, which is related to the maximum speed, strength and explosive force of the lower limbs. For this test, participants stood on the Kistler force measurement platform (9260AA, Kistler Co., Ltd., Switzerland) on both feet and performed to inspection. During the test, they were asked to put their hands on their hips and remain on the platform. After that, they were asked to squat down until the knees bent 90 degrees and then to immediately jump as high as possible. The strength development speed (30 ms) were recorded during the jump. Each participant repeated the test 3 times, and CMJ data were obtained at the designated points. The instrument was calibrated for each individual's weight.
Wingate Anaerobic Test (WAnT) | From Baseline to 6 Weeks Assessed
  After a standard warm-up, all subjects were assessed with the classical WAnT on a cycloergometer (Monark 894E, Varberg, Sweden) in a 30 s "go all out" ultramax test. The seat height was adjusted to the satisfaction of each participant, and toe clips prevented the feet from slipping off the pedals. Before the initial test, the subjects warmed up for 5 min, and the power was approximately 50 W. After the warm-up, two preparation exercises lasting 3 s, during which the actual test load was 3% of their own body weight, were applied to accustom the participant to resistance. The test started, and the resistance was set on the friction belt of the dynamometer. External loading was estimated individually at 5% body weight. The recorded results were the relative mean power (W/kg), relative peak power (W/kg), and fatigue index (%). This assessment was performed before and 24 and 72 h after the exhaustive exercise program.
Isometric Mid-Thigh Pull (IMTP) | From Baseline to 6 Weeks Assessed
  Customized IMTP test equipment and two force plates (type 9287BA, Kistler Instruments AG, Winterthur, Switzerland) were used. All participants stood with their feet the same width apart, and the rod was placed between the thighs, with the torso upright, the spine neutral, and the knee and hip angles at 140°, to familiarize the participants with the IMPT test method. The average absolute peak force (PF), relative peak force (N/Kg), rate of force development (RFD), peak rate of force development (pRFD), time to peak force (TPF) and time to peak rate of force development (TPRFD) parameters were recorded. This assessment was performed before and 24 and 48h after the exhaustive exercise program.
Isometric Mid-Thigh Pull (IMTP) | From Baseline to 6 Weeks Assessed. This assessment was performed before and 24 and 48h after the exhaustive exercise program.
  Customized IMTP test equipment and two force plates (type 9287BA, Kistler Instruments AG, Winterthur, Switzerland) were used. All participants stood with their feet the same width apart, and the rod was placed between the thighs, with the torso upright, the spine neutral, and the knee and hip angles at 140°, to familiarize the participants with the IMPT test method. The average absolute peak force (PF) were recorded.
Isometric Mid-Thigh Pull (IMTP) | From Baseline to 6 Weeks Assessed. This assessment was performed before and 24 and 48h after the exhaustive exercise program.
  Customized IMTP test equipment and two force plates (type 9287BA, Kistler Instruments AG, Winterthur, Switzerland) were used. All participants stood with their feet the same width apart, and the rod was placed between the thighs, with the torso upright, the spine neutral, and the knee and hip angles at 140°, to familiarize the participants with the IMPT test method. The average absolute peak rate of force development (RFD) parameters were recorded.

SECONDARY OUTCOMES:
Gut microbiota | From Baseline to 6 Weeks Assessed
  Collect the DNA of fecal flora to test the diversity and abundance of gut microbiota in Stool samples before and after probiotics
Change in Perceived Stress Scale (PSS) Score From Baseline to Change in Perceived Stress Scale (PSS) | From Baseline to 6 Weeks Assessed
  The PSS scores is a rating tool used to gauge the course of stree. The minimum total score possible is 0 and the maximum total score possible is 40. Higher values represent a worse outcome.
Differences in the The Profile of Mood States (POMS) before and after probiotics consumption | From Baseline to 6 Weeks Assessed
  The Profile of Mood States (POMS) is a psychological rating scale used to assess transient, distinct mood states. The Chinese version POMS measures six different dimensions of mood swings over a period of time. These include: Tension or Anxiety, Anger or Hostility, Vigor or Activity, Fatigue or Inertia, Depression or Dejection, Confusion or Bewilderment. A four-point scale ranging from "not at all" to "extremely" is administered by experimenters to patients to assess their mood states.
The Quality of Life, Enjoyment, and Satisfaction Questionnaire-16, QLESQ-16 | From Baseline to 6 Weeks Assessed
  The Quality of Life, Enjoyment, and Satisfaction Questionnaire-16 (QLESQ-16) is a valid, reliable self-report instrument for assessing quality of life.
Visual Analogue Scale-GI (VAS-GI) | From Baseline to 6 Weeks Assessed
  Visual Analogue Scale (VAS) consists of a line, 10 cm in length. Individuals point to or mark a spot on the line where they feel indicates their current their emotion, fatigue level and sleep quality. The score of emotion level is from 0cm (very nervous) to 10 cm (very relaxing). The score of fatigue level is from 0 cm (very energetic) to 10 cm (very sleepy). The score of sleep quality is from 0 cm (poor) to 10 cm (sleep well). The maximum total score is 100% (equal 10cm).
Change in Patient Global Impression of Change (PGIC) | From Baseline to 6 Weeks Assessed
  The PGIC consists of one item taken from the clinical global impression and adapted to the patient. The minimum total score possible is 1 and the maximum total score possible is 7. Higher values represent a worse outcome.
Safety assessment - AST | From Baseline to 6 Weeks Assessed
  Safety is assessed function of liver and kidney such as AST (8-38 IU/L).
Safety assessment - ALT | From Baseline to 6 Weeks Assessed
  Safety is assessed function of liver and kidney such as ALT (4-44 IU/L).
Safety assessment - T-Cholesterol | From Baseline to 6 Weeks Assessed
  Safety is assessed function of liver and kidney such as T-Cholesterol (<170 mg/dL).
Safety assessment - Uric Acid | From Baseline to 6 Weeks Assessed
  Safety is assessed function of liver and kidney such as Uric Acid (3.4-7.6 mg/dl)
Safety assessment - Bun | From Baseline to 6 Weeks Assessed
  Safety is assessed function of liver and kidney such as Bun (6-20 mg/dl)
Safety assessment - Creatinine | From Baseline to 6 Weeks Assessed
  Safety is assessed function of liver and kidney such as Creatinine (0.6-1.3 mg/dl)
Safety assessment - Glucose | From one week before Baseline to 6 Weeks Assessed
  Safety is assessed function of liver and kidney such as Glucose (70~100 mg/dL)
Safety assessment - Triglycerides | From Baseline to 6 Weeks Assessed
  Safety is assessed function of liver and kidney such as Triglycerides (<150 mg/dL)
Safety assessment - LDL | From Baseline to 6 Weeks Assessed
  Safety is assessed function of liver and kidney such as LDL (0~140mg/dl)
Safety assessment - HDL | From Baseline to 6 Weeks Assessed
  Safety is assessed function of liver and kidney such as HDL (>40mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Chang Huang, Ph.D, Principal Investigator — National Taiwan Sport University
Locations (1):
- National Taiwan Sport University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided